CLINICAL TRIAL: NCT04113876
Title: Circadian Health in Patients Admitted to Intensive Care Units and Hospitalization (CHRONOHOSPI)
Brief Title: Circadian Health and Influential Factors
Acronym: CHRONOHOSPI
Status: Completed | Type: Observational
Sponsor: Instituto de Salud Carlos III (Other Government)
Collaborators: Institut de Recerca Biomèdica de Lleida (Other); Instituto Murciano de Investigación Biosanitaria Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Teresa Moreno Casbas, Doctor, Clinical Research, Instituto de Salud Carlos III
Other Study IDs: PI18/2019-v3
Record Dates: First submitted 2019-09-06; First posted 2019-10-03 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Chronobiology Disorders
Keywords: sleep quality; circadian rhythm; nursing activities
MeSH Terms: conditions — Chronobiology Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the quality of sleep of patients admitted to medical and intensive care units. All of them will have a clock placed to measure their circadian activity. Also, data will be recorded through questionnaires about the unit, patient habits and medical problems.

DETAILED DESCRIPTION:
The investigators found an extensive bibliography related to the quality of sleep and its effects on health. However, it should be noted the literary emptiness in relation to the influential factors in it. Chronobiology is the science responsible for studying the rhythmic changes in living beings; where the investigators include the circadian rhythm. In this way, all the "cycles" will be influenced by a series of factors that allow its correct operation, being in this case the light-dark cycle (LD), together with the temperature compensation, these being the determinants that allow, or not homeostasis.

The sleep - wake pattern is one of the most important circadian rhythms that happen in the organism. The dream is an unconscious process by which, despite the muscular relaxation that occurs, it is accompanied by continuous brain activity along with sensitive perception, where several of the organ systems come into play. This cycle is composed of two factors: a homeostatic one directly proportional to the time we are awake, and another circadian, dependent on the secretion of melatonin and the body's regulation of temperature. This fact can be compromised by the appearance of both external and internal stimuli, altering normal functioning, which is translated into sleep deprivation, which, if extended over time, can have physical and mental consequences, Some of them are: deterioration of the immune function, an increase in the incidence of cardiovascular diseases, memory deficit, early aging, mood swings, difficulty in healing, greater probability of developing metabolic syndromes, cognitive, affective disorders and even some types of cancer

The results obtained will facilitate the elaboration of action protocols focused on improving sleep quality in hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* subjects over 18 years of age, minimum duration of the hospitalization process of 96h, conscious and oriented with constancy in their clinical history (HC) and who give their consent.

Exclusion Criteria:

* personas con discapacidad visual y/o auditiva documentada en su HC, en el caso de los pacientes de Unidades de Cuidados Intensivos (UCIs) se excluirán a aquellos que obtengan una puntuación inferior a 8 en la escala Glasgow. Pacientes con cualquier tipo de aislamiento y aquellos incluidos en el plan de Cuidados Paliativos.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Users who are part of the study must be adults admitted to intensive care units (ICUs), Medical Units (UMs) and Surgical units (UQs), of the 13 participating hospitals: Andalusia (H. Juan Ramón Jiménez, Huelva), Catalonia (H. Mataró and H. Arnau Villanova, Lleida), Cantabria (HU Marqués Valdecilla), Castilla y León (H. del Bierzo, Ponferrada), Castila-La Mancha (HGU Ciudad Real), C. Madrid (HU 12 de Octubre ), C. Valenciana (HGU Valencia and HGU Alicante), Murcia Region (C H Cartagena, HCU V Arrixaca) and Basque Country (H. Basurto, Bilbao and H. Galdakao-Usansolo, Vizcaya).
Sampling Method: Non-Probability Sample
Enrollment: 975 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Circadian Health | 96 hours
  Using the KRONOHEALTH® recording device, we will measure the following indicators:
  * Total Sleep Time
  * Sleep Fragmentations
  * Sleep depth
  * Chronobiological health index

SECONDARY OUTCOMES:
Subjective Sleep Quality | 1 day (one time evaluation)
  Scores in the Pittsburgh sleep quality index
Degree of sleep interference during hospitalization | 1 day (one time evaluation)
  Visual analogue scale from 0 to 10 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Teresa Moreno Casbas, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Erren TC, Reiter RJ. Revisiting chronodisruption: when the physiological nexus between internal and external times splits in humans. Naturwissenschaften. 2013 Apr;100(4):291-8. doi: 10.1007/s00114-013-1026-5. Epub 2013 Mar 14. PMID 23494200
- [Result] Erren TC, Reiter RJ. Defining chronodisruption. J Pineal Res. 2009 Apr;46(3):245-7. doi: 10.1111/j.1600-079X.2009.00665.x. Epub 2009 Feb 9. PMID 19215573
- [Result] Garaulet M, Madrid JA. Chronobiological aspects of nutrition, metabolic syndrome and obesity. Adv Drug Deliv Rev. 2010 Jul 31;62(9-10):967-78. doi: 10.1016/j.addr.2010.05.005. Epub 2010 May 24. PMID 20580916
- [Result] Saper CB, Scammell TE, Lu J. Hypothalamic regulation of sleep and circadian rhythms. Nature. 2005 Oct 27;437(7063):1257-63. doi: 10.1038/nature04284. PMID 16251950
- [Result] Tononi G, Cirelli C. Sleep function and synaptic homeostasis. Sleep Med Rev. 2006 Feb;10(1):49-62. doi: 10.1016/j.smrv.2005.05.002. Epub 2005 Dec 22. PMID 16376591
- [Result] Martínez Nicolás AB, Blázquez Manzanera A. La hora de nuestro cuerpo. Monitorización Ambulatoria Circadiana. Revista Eubacteria 2015; 33: 22-28.
- [Result] 8 National Institute of Neurological Disorders and Stroke. (2007). How much sleep do we need? In Brain Basics: Understanding Sleep. [obtenido de: http://bit.ly/2rA34Zk consultado 30 de enero de 2018].
- [Result] da Costa SV, Ceolim MF. [Factors that affect inpatients' quality of sleep]. Rev Esc Enferm USP. 2013 Feb;47(1):46-52. doi: 10.1590/s0080-62342013000100006. Portuguese. PMID 23515802
- [Result] Hacker ED, Kapella MC, Park C, Ferrans CE, Larson JL. Sleep Patterns During Hospitalization Following Hematopoietic Stem Cell Transplantation. Oncol Nurs Forum. 2015 Jul;42(4):371-9. doi: 10.1188/15.ONF.371-379. PMID 26148316
- [Result] Van Someren EJ, Cirelli C, Dijk DJ, Van Cauter E, Schwartz S, Chee MW. Disrupted Sleep: From Molecules to Cognition. J Neurosci. 2015 Oct 14;35(41):13889-95. doi: 10.1523/JNEUROSCI.2592-15.2015. PMID 26468189
- [Result] Cho K, Ennaceur A, Cole JC, Suh CK. Chronic jet lag produces cognitive deficits. J Neurosci. 2000 Mar 15;20(6):RC66. doi: 10.1523/JNEUROSCI.20-06-j0005.2000. PMID 10704520
- [Result] Pandi-Perumal SR, Moscovitch A, Srinivasan V, Spence DW, Cardinali DP, Brown GM. Bidirectional communication between sleep and circadian rhythms and its implications for depression: lessons from agomelatine. Prog Neurobiol. 2009 Aug;88(4):264-71. doi: 10.1016/j.pneurobio.2009.04.007. Epub 2009 May 18. PMID 19454302
- [Result] Davis S, Mirick DK, Stevens RG. Night shift work, light at night, and risk of breast cancer. J Natl Cancer Inst. 2001 Oct 17;93(20):1557-62. doi: 10.1093/jnci/93.20.1557. PMID 11604479
- [Result] Kondratov RV. A role of the circadian system and circadian proteins in aging. Ageing Res Rev. 2007 May;6(1):12-27. doi: 10.1016/j.arr.2007.02.003. Epub 2007 Feb 21. PMID 17369106
- [Result] Venkateshiah SB, Collop NA. Sleep and sleep disorders in the hospital. Chest. 2012 May;141(5):1337-1345. doi: 10.1378/chest.11-2591. PMID 22553268
- [Result] Young JS, Bourgeois JA, Hilty DM, Hardin KA. Sleep in hospitalized medical patients, part 1: factors affecting sleep. J Hosp Med. 2008 Nov-Dec;3(6):473-82. doi: 10.1002/jhm.372. PMID 19084897
- [Result] Erren TC, Reiter RJ. Preventing cancers caused by chronodisruption: blocking blue light alone is unlikely to do the trick. Med Hypotheses. 2009 Dec;73(6):1077-8. doi: 10.1016/j.mehy.2009.05.003. Epub 2009 Jun 3. No abstract available. PMID 19497681
- [Result] Portas CM, Krakow K, Allen P, Josephs O, Armony JL, Frith CD. Auditory processing across the sleep-wake cycle: simultaneous EEG and fMRI monitoring in humans. Neuron. 2000 Dec;28(3):991-9. doi: 10.1016/s0896-6273(00)00169-0. PMID 11163282
- [Result] Halperin D. Environmental noise and sleep disturbances: A threat to health? Sleep Sci. 2014 Dec;7(4):209-12. doi: 10.1016/j.slsci.2014.11.003. Epub 2014 Nov 15. PMID 26483931
- [Result] Delaney LJ, Van Haren F, Lopez V. Sleeping on a problem: the impact of sleep disturbance on intensive care patients - a clinical review. Ann Intensive Care. 2015 Feb 26;5:3. doi: 10.1186/s13613-015-0043-2. eCollection 2015. PMID 25852963
- [Result] Little A, Ethier C, Ayas N, Thanachayanont T, Jiang D, Mehta S. A patient survey of sleep quality in the Intensive Care Unit. Minerva Anestesiol. 2012 Apr;78(4):406-14. Epub 2012 Feb 15. PMID 22337154
- [Result] Carvalho Bos S, Waterhouse J, Edwards B, Simons R, Reilly T. The use of actimetry to assess changes to the rest-activity cycle. Chronobiol Int. 2003 Nov;20(6):1039-59. doi: 10.1081/cbi-120025397. PMID 14680142
- [Result] Roenneberg T, Kuehnle T, Juda M, Kantermann T, Allebrandt K, Gordijn M, Merrow M. Epidemiology of the human circadian clock. Sleep Med Rev. 2007 Dec;11(6):429-38. doi: 10.1016/j.smrv.2007.07.005. Epub 2007 Nov 1. PMID 17936039
- [Result] Ancoli-Israel S, Cole R, Alessi C, Chambers M, Moorcroft W, Pollak CP. The role of actigraphy in the study of sleep and circadian rhythms. Sleep. 2003 May 1;26(3):342-92. doi: 10.1093/sleep/26.3.342. PMID 12749557
- [Result] Morgenthaler T, Alessi C, Friedman L, Owens J, Kapur V, Boehlecke B, Brown T, Chesson A Jr, Coleman J, Lee-Chiong T, Pancer J, Swick TJ; Standards of Practice Committee; American Academy of Sleep Medicine. Practice parameters for the use of actigraphy in the assessment of sleep and sleep disorders: an update for 2007. Sleep. 2007 Apr;30(4):519-29. doi: 10.1093/sleep/30.4.519. PMID 17520797
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888